CLINICAL TRIAL: NCT01135758
Title: Pilot Study Probing the Antidepressant Effects of 0.5 mg/kg Intravenous Ketamine in Drug-resistant Depressed Patients (Unipolar Depression): Efficacy, Safety, Brain Function
Brief Title: Study of Depression-Ketamine-Brain Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of funding of study
Sponsor: Markus KOSEL (Other)
Responsible Party: Sponsor-Investigator, Markus KOSEL, MD-PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE09-144/Psy 09-22
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Major Depression
Keywords: depression, ketamine, fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ketamine 0.5 mg/kg i.v. (Experimental): Single administration of ketamine 0.5 mg/kg i.v.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Administration of a subanaesthetic dose of Ketamine, intravenously (0.5 mg/kg)

SUMMARY:
Targeting the glutamatergic system to treat depression is a new and promising strategy based on studies at the molecular, synaptic, and neuronal level but also on results of studies conducted in animal models and first clinical studies involving depressed patients.Ketamine has been proposed as a novel approach to induce rapid antidepressant response. In this pilot project the investigators aim to introduce this novel and promising approach into clinical practice. Besides the assessment of clinical efficacy, the investigators will put a special emphasis on the assessment of ketamine-associated effects on brain function using fMRI and cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years with a diagnosis of major depressive disorder without psychotic features.
* Drug-resistant depressed patients (defined as non-response to two sufficiently long (at least 6 weeks) drug trials at the maximal authorized or tolerated dose)
* Score 25 or higher on the Montgomery-Asberg Depression Rating Scale
* Stable psychotropic medication (antidepressants, antipsychotics, mood stabilizers) during the last 6 weeks prior to inclusion.
* Legally competent subjects agreeing to comply with the requirements of the study and authorizing the transmission of relevant information to competent physicians in the case of a clinically relevant previously unknown finding during an MRI examination.

Exclusion Criteria:

* Subjects with co-morbid substance abuse or dependence during the 3 months prior to inclusion, except nicotine consumption.
* Patients judged to be at serious suicide risk (score ≥ 4 at item 10 of the MADRS).
* Patients with any other DSM-IV axis one diagnosis including bipolar disorder except for anxiety disorder which are not dominating the clinical presentation.
* History of antidepressant or substance-induced hypomania or mania.
* History of psychotic symptoms.
* Patients with any contra-indication to the administration of ketamine, especially present diagnosis or antecedents of clinically relevant cardiovascular disorders (clinically significant or not adequately treated hypertension, present or previous diagnosis of cardiovascular disorder such as stroke or heart attack etc).
* Any MRI contraindication, especially metallic implants, pacemaker, etc.
* Pregnant women, breast-feeding women, women of childbearing age without effective means of contraception.
* Treatment during the last 2 weeks with thyroid hormones and sympathicomimetic drug.
* Present or past diagnosis of eclampsia or preeclampsia.
* Untreated or insufficiently treated hyperthyroidism.
* Known hypersensitivity to ketamine or to the excipient (benzethonium chloride).
* Present or past diagnosis of glaucoma, intracranial hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference of the MADRS score at baseline and after ketamine injection | 40, 80, 110, 230 min, 1, 2, 3, 6, 7, 10 d after ketamine administration

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kosel, MD-PhD, Principal Investigator — Departement of Adult Psychiatry, University Hospital of Geneva
Locations (1):
- Service de Psychiatrie Adulte, Programme dépression, Geneva, Switzerland